CLINICAL TRIAL: NCT00180271
Title: Multicenter Automatic Defibrillator Implantation Trial With Cardiac Resynchronization Therapy
Brief Title: MADIT-CRT: Multicenter Automatic Defibrillator Implantation With Cardiac Resynchronization Therapy
Acronym: MADIT-CRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: University of Rochester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Clinicals0003; MADIT-CRT
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Results first posted 2011-06-02 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Tachycardia; Congestive Heart Failure
Keywords: Defibrillator; Cardiac Resynchronization Therapy; MADIT
MeSH Terms: conditions — Tachycardia; Heart Failure | interventions — Cardiac Resynchronization Therapy; Electric Countershock; Defibrillators, Implantable

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CRT-D (Experimental): CRT-D: Cardiac resynchronization therapy with defibrillation.
  Interventions: Device: Cardiac resynchronization therapy with defibrillation
- ICD (Active Comparator): ICD: Implantable cardioverter defibrillator
  Interventions: Device: Implantable Cardioverter Defibrillator (ICD)

INTERVENTIONS:
Device: Cardiac resynchronization therapy with defibrillation — Boston Scientific Corporation Market Released Cardiac Resynchronization therapy with defibrillation
  Arms: CRT-D
Device: Implantable Cardioverter Defibrillator (ICD) — Boston Scientific Corporation Market Released Implantable Cardioverter Defibrillator
  Arms: ICD

SUMMARY:
The MADIT-CRT trial is designed to determine if combined implantable cardiac defibrillator (ICD)-cardiac resynchronization therapy (CRT-D) will reduce the risk of mortality and heart failure (HF) events by approximately 25%, in subjects who are in New York Heart Association (NYHA) functional Class II with non-ischemic or ischemic cardiomyopathy and subjects who are in NYHA functional Class I with ischemic cardiomyopathy, left ventricular dysfunction (ejection fraction [EF] < or = 0.30), and prolonged intraventricular conduction (QRS duration > or = 130 ms).

DETAILED DESCRIPTION:
In this study, subjects will be randomized to CRT-D or ICD-only. Randomization will be stratified by clinical center and ischemic status. Approximately 60% of the subjects will be randomly assigned to receive a CRT-D with biventricular pacing, and 40% will receive an ICD only. Optimal pharmacological therapy for heart failure will be required in both treatment arms. Length of follow-up for each subject will depend on the date of entry into the study, since all subjects will be followed to a common study termination date.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic heart disease defined as:

  * NYHA Class I or II for the past 3 calendar months prior to, and at the time of, enrollment;
  * one or more clinically documented (Q wave or enzyme positive) prior myocardial infarctions, but not within 3 calendar months of enrollment; and/or
  * one or more prior coronary artery bypass graft surgeries or percutaneous coronary interventions (balloon and/or stent angioplasty) but not within 3 calendar months of enrollment.

OR

* Non-ischemic heart disease including dilated cardiomyopathy characterized by a low ejection fraction and increased ventricular volume, with ventricular compliance that is normal or increased
* NYHA Class II for the past 3 calendar months prior to, and at the time of, enrollment

AND all of the following:

* Stable optimal pharmacologic therapy.
* An ejection fraction < or = 0.30 by angiographic, radionuclide, or echocardiographic methods within one year prior to enrollment and measured during the enrollment echocardiogram obtained within 14 days prior to randomization to confirm eligibility (recommended)
* Resting QRS duration > or = 130 ms on print-out of a current electrocardiogram (ECG) obtained within 14 days prior to randomization.
* Sinus rhythm by ECG (including right bundle branch block [RBBB] and first degree heart block with PR < 250 ms.)
* Men and women 21 years of age or older (no upper-age cut off)

Exclusion Criteria:

* Existing indication for CRT
* Subjects with an implanted pacemaker
* Subjects with an existing ICD or CRT device
* Subjects in NYHA Class I with non-ischemic cardiomyopathy
* Subjects in NYHA Class III or IV in the past 3 calendar months prior to, or at the time of, enrollment
* Coronary artery bypass graft surgery or percutaneous coronary intervention (balloon and/or stent angioplasty) within the past 3 calendar months prior to enrollment
* Enzyme-positive myocardial infarction within the past 3 calendar months prior to enrollment
* Subjects with angiographic evidence of coronary disease who are candidates for coronary revascularization and are likely to undergo coronary artery bypass graft surgery or percutaneous coronary intervention in the foreseeable future
* Subjects with second or third degree heart block
* Subjects with irreversible brain damage from preexisting cerebral disease
* Women who are pregnant or plan to become pregnant during the course of the trial. Women of childbearing potential must have a negative pregnancy test within 7 days prior to enrollment.
* Reversible non-ischemic cardiomyopathy such as acute viral myocarditis or discontinuation of alcohol in alcohol-induced heart disease
* Subjects with chronic atrial fibrillation within one month prior to enrollment
* Presence of any disease, other than the subject's cardiac disease, associated with a reduced likelihood of survival for the duration of the trial, e.g., cancer, uremia (blood urea nitrogen [BUN] > 70 mg/dl or creatinine > 3.0 mg/dl), liver failure, etc.
* Subjects participating in any other clinical trials
* Subjects unwilling or unable to cooperate with the protocol
* Subjects who live at such a distance from the clinic that travel for follow-up visits would be unusually difficult
* Subjects who do not anticipate being residents of the area for the scheduled duration of the trial
* Subjects unwilling to sign the consent for participation

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1820 (Actual)
Dates: Start 2004-12; Primary Completion 2009-06 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur J Moss, MD, Principal Investigator — University of Rochester, NY
Locations (1):
- Multiple locations in the US and international, Rochester, New York, United States

REFERENCES:
- [Derived] Fudim M, Dalgaard F, Friedman DJ, Abraham WT, Cleland JGF, Curtis AB, Gold MR, Kutyifa V, Linde C, Ali-Ahmed F, Tang A, Olivas-Martinez A, Inoue LYT, Al-Khatib SM, Sanders GD. Comorbidities and clinical response to cardiac resynchronization therapy: Patient-level meta-analysis from eight clinical trials. Eur J Heart Fail. 2024 Apr;26(4):1039-1046. doi: 10.1002/ejhf.3029. Epub 2023 Sep 15. PMID 37671601
- [Derived] Friedman DJ, Al-Khatib SM, Dalgaard F, Fudim M, Abraham WT, Cleland JGF, Curtis AB, Gold MR, Kutyifa V, Linde C, Tang AS, Ali-Ahmed F, Olivas-Martinez A, Inoue LYT, Sanders GD. Cardiac Resynchronization Therapy Improves Outcomes in Patients With Intraventricular Conduction Delay But Not Right Bundle Branch Block: A Patient-Level Meta-Analysis of Randomized Controlled Trials. Circulation. 2023 Mar 7;147(10):812-823. doi: 10.1161/CIRCULATIONAHA.122.062124. Epub 2023 Jan 26. PMID 36700426
- [Derived] Goldenberg I, Younis A, Aktas MK, McNitt S, Zareba W, Kutyifa V. Competing risk analysis of ventricular arrhythmia events in heart failure patients with moderately compromised renal dysfunction. Europace. 2020 Sep 1;22(9):1384-1390. doi: 10.1093/europace/euaa146. PMID 32875313
- [Derived] Younis A, Goldenberg M, Kutyifa V, Polonsky B, Mcnitt S, Zareba W, Golovchiner G, Aktas MK, Barsheshet A. Applicability of the MADIT-CRT Response Score for Prediction of Long-Term Clinical and Arrhythmic Events by QRS Morphology. Circ Arrhythm Electrophysiol. 2020 Sep;13(9):e008499. doi: 10.1161/CIRCEP.120.008499. Epub 2020 Jul 23. No abstract available. PMID 32701367
- [Derived] Vidula H, Lee E, McNitt S, Polonsky B, Aktas M, Rosero S, Younis A, Solomon SD, Zareba W, Kutyifa V, Goldenberg I. Cardiac Resynchronization Therapy and Risk of Recurrent Hospitalizations in Patients Without Left Bundle Branch Block: The Long-Term Multicenter Automatic Defibrillator Implantation Trial With Cardiac Resynchronization Therapy. Circ Heart Fail. 2020 Jul;13(7):e006925. doi: 10.1161/CIRCHEARTFAILURE.120.006925. Epub 2020 Jul 1. PMID 32605387
- [Derived] Biton Y, Daimee UA, Baman JR, Kutyifa V, McNitt S, Polonsky B, Zareba W, Goldenberg I. Prognostic Importance of Defibrillator-Appropriate Shocks and Antitachycardia Pacing in Patients With Mild Heart Failure. J Am Heart Assoc. 2019 Mar 19;8(6):e010346. doi: 10.1161/JAHA.118.010346. PMID 30857452
- [Derived] Kutyifa V, Vermilye K, Solomon SD, McNitt S, Moss AJ, Daimee UA. Long-term outcomes of cardiac resynchronization therapy by left ventricular ejection fraction. Eur J Heart Fail. 2019 Mar;21(3):360-369. doi: 10.1002/ejhf.1357. Epub 2018 Dec 28. PMID 30592353
- [Derived] Baturova MA, Kutyifa V, McNitt S, Polonsky B, Solomon S, Carlson J, Zareba W, Platonov PG. Usefulness of Electrocardiographic Left Atrial Abnormality to Predict Response to Cardiac Resynchronization Therapy in Patients With Mild Heart Failure and Left Bundle Branch Block (a Multicenter Automatic Defibrillator Implantation Trial with Cardiac Resynchronization Therapy Substudy). Am J Cardiol. 2018 Jul 15;122(2):268-274. doi: 10.1016/j.amjcard.2018.03.364. Epub 2018 Apr 11. PMID 29861050
- [Derived] Ozlu MF, Barsheshet A, Moss AJ, Goldenberg I, Kutyifa V, Biton Y, McNitt S, Zareba W, Aktas MK. Time Dependence of Ventricular Tachyarrhythmias After Myocardial Infarction: A MADIT-CRT Substudy. JACC Clin Electrophysiol. 2016 Oct;2(5):565-573. doi: 10.1016/j.jacep.2016.04.010. Epub 2016 Jun 22. PMID 29759576
- [Derived] Jame S, Kutyifa V, Polonsky B, McNitt S, Al-Ahmad A, Moss AJ, Zareba W, Wang PJ. Predictive value of device-derived activity level for short-term outcomes in MADIT-CRT. Heart Rhythm. 2017 Jul;14(7):1081-1086. doi: 10.1016/j.hrthm.2017.03.032. Epub 2017 Mar 25. PMID 28347835
- [Derived] Biering-Sorensen T, Knappe D, Pouleur AC, Claggett B, Wang PJ, Moss AJ, Solomon SD, Kutyifa V. Regional Longitudinal Deformation Improves Prediction of Ventricular Tachyarrhythmias in Patients With Heart Failure With Reduced Ejection Fraction: A MADIT-CRT Substudy (Multicenter Automatic Defibrillator Implantation Trial-Cardiac Resynchronization Therapy). Circ Cardiovasc Imaging. 2017 Jan;10(1):e005096. doi: 10.1161/CIRCIMAGING.116.005096. PMID 28003221
- [Derived] Mathias A, Moss AJ, McNitt S, Zareba W, Goldenberg I, Solomon SD, Kutyifa V. Clinical Implications of Complete Left-Sided Reverse Remodeling With Cardiac Resynchronization Therapy: A MADIT-CRT Substudy. J Am Coll Cardiol. 2016 Sep 20;68(12):1268-76. doi: 10.1016/j.jacc.2016.06.051. PMID 27634117
- [Derived] Jame S, Kutyifa V, Aktas MK, McNitt S, Polonsky B, Al-Ahmad A, Zareba W, Moss A, Wang PJ. Bipolar left ventricular pacing is associated with significant reduction in heart failure or death in CRT-D patients with LBBB. Heart Rhythm. 2016 Jul;13(7):1468-74. doi: 10.1016/j.hrthm.2016.03.009. Epub 2016 Mar 4. PMID 26961303
- [Derived] Biton Y, Kutyifa V, Cygankiewicz I, Goldenberg I, Klein H, McNitt S, Polonsky B, Ruwald AC, Ruwald MH, Moss AJ, Zareba W. Relation of QRS Duration to Clinical Benefit of Cardiac Resynchronization Therapy in Mild Heart Failure Patients Without Left Bundle Branch Block: The Multicenter Automatic Defibrillator Implantation Trial with Cardiac Resynchronization Therapy Substudy. Circ Heart Fail. 2016 Feb;9(2):e002667. doi: 10.1161/CIRCHEARTFAILURE.115.002667. PMID 26823498
- [Derived] Biton Y, Goldenberg I, Kutyifa V, Baman JR, Solomon S, Moss AJ, Szepietowska B, McNitt S, Polonsky B, Zareba W, Barsheshet A. Relative Wall Thickness and the Risk for Ventricular Tachyarrhythmias in Patients With Left Ventricular Dysfunction. J Am Coll Cardiol. 2016 Jan 26;67(3):303-12. doi: 10.1016/j.jacc.2015.10.076. PMID 26796396
- [Derived] Medina A, Moss AJ, McNitt S, Zareba W, Wang PJ, Goldenberg I. Brain natriuretic peptide and the risk of ventricular tachyarrhythmias in mildly symptomatic heart failure patients enrolled in MADIT-CRT. Heart Rhythm. 2016 Apr;13(4):852-9. doi: 10.1016/j.hrthm.2015.12.024. Epub 2015 Dec 25. PMID 26724489
- [Derived] Biton Y, Goldenberg I, Kutyifa V, Zareba W, Szepietowska B, Mcnitt S, Polonsky B, Barsheshet A, Moss AJ. Effects of Statins on First and Recurrent Supraventricular Arrhythmias in Patients With Mild Heart Failure (from the Multicenter Automatic Defibrillator Implantation Trial With Cardiac Resynchronization Therapy). Am J Cardiol. 2015 Dec 15;116(12):1869-74. doi: 10.1016/j.amjcard.2015.09.027. Epub 2015 Oct 8. PMID 26508711
- [Derived] Biton Y, Kutyifa V, Zareba W, Klein HU, Solomon SD, McNitt S, Polonsky B, Moss AJ, Goldenberg I. Long-term outcome with cardiac resynchronization therapy in mild heart failure patients with left bundle branch block from US and Europe MADIT-CRT. Heart Fail Rev. 2015 Sep;20(5):535-43. doi: 10.1007/s10741-015-9499-2. PMID 26216033
- [Derived] Biton Y, Moss AJ, Kutyifa V, Mathias A, Sherazi S, Zareba W, McNitt S, Polonsky B, Barsheshet A, Brown MW, Goldenberg I. Inverse Relationship of Blood Pressure to Long-Term Outcomes and Benefit of Cardiac Resynchronization Therapy in Patients With Mild Heart Failure: A Multicenter Automatic Defibrillator Implantation Trial With Cardiac Resynchronization Therapy Long-Term Follow-Up Substudy. Circ Heart Fail. 2015 Sep;8(5):921-6. doi: 10.1161/CIRCHEARTFAILURE.115.002208. Epub 2015 Jul 15. PMID 26179186
- [Derived] Kutyifa V, Moss AJ, Solomon SD, McNitt S, Aktas MK, Barsheshet A, Merkely B, Zareba W, Goldenberg I. Reduced risk of life-threatening ventricular tachyarrhythmias with cardiac resynchronization therapy: relationship to left ventricular ejection fraction. Eur J Heart Fail. 2015 Sep;17(9):971-8. doi: 10.1002/ejhf.311. Epub 2015 Jul 14. PMID 26173635
- [Derived] Biton Y, Zareba W, Goldenberg I, Klein H, McNitt S, Polonsky B, Moss AJ, Kutyifa V; MADIT-CRT Executive Committee. Sex Differences in Long-Term Outcomes With Cardiac Resynchronization Therapy in Mild Heart Failure Patients With Left Bundle Branch Block. J Am Heart Assoc. 2015 Jun 29;4(7):e002013. doi: 10.1161/JAHA.115.002013. PMID 26124205
- [Derived] Perkiomaki JS, Ruwald AC, Kutyifa V, Ruwald MH, Mcnitt S, Polonsky B, Goldstein RE, Haigney MC, Krone RJ, Zareba W, Moss AJ; MADIT-CRT Investigators. Risk factors and the effect of cardiac resynchronization therapy on cardiac and non-cardiac mortality in MADIT-CRT. Europace. 2015 Dec;17(12):1816-22. doi: 10.1093/europace/euv201. Epub 2015 Jun 11. PMID 26071234
- [Derived] Daimee UA, Moss AJ, Biton Y, Solomon SD, Klein HU, McNitt S, Polonsky B, Zareba W, Goldenberg I, Kutyifa V. Long-Term Outcomes With Cardiac Resynchronization Therapy in Patients With Mild Heart Failure With Moderate Renal Dysfunction. Circ Heart Fail. 2015 Jul;8(4):725-32. doi: 10.1161/CIRCHEARTFAILURE.115.002082. Epub 2015 Jun 2. PMID 26038537
- [Derived] Lee AY, Moss AJ, Ruwald MH, Kutyifa V, McNitt S, Polonsky B, Zareba W, Ruwald AC. Temporal Influence of Heart Failure Hospitalizations Prior to Implantable Cardioverter Defibrillator or Cardiac Resynchronization Therapy With Defibrillator on Subsequent Outcome in Mild Heart Failure Patients (from MADIT-CRT). Am J Cardiol. 2015 May 15;115(10):1423-7. doi: 10.1016/j.amjcard.2015.02.029. Epub 2015 Feb 18. PMID 25817576
- [Derived] Aktas MK, Goldenberg I, Moss AJ, Huang DT, Kutyifa V, Wang PJ, Brenyo A, McNitt S, Zareba W, Barsheshet A. Comparison of age (<75 Years versus >/=75 Years) to risk of ventricular tachyarrhythmias and implantable cardioverter defibrillator shocks (from the Multicenter Automatic Defibrillator Implantation Trial With Cardiac Resynchronization Therapy). Am J Cardiol. 2014 Dec 15;114(12):1855-60. doi: 10.1016/j.amjcard.2014.09.026. Epub 2014 Sep 28. PMID 25438913
- [Derived] Ruwald MH, Moss AJ, Zareba W, Jons C, Ruwald AC, McNitt S, Polonsky B, Kutyifa V. Circadian distribution of ventricular tachyarrhythmias and association with mortality in the MADIT-CRT trial. J Cardiovasc Electrophysiol. 2015 Mar;26(3):291-9. doi: 10.1111/jce.12592. Epub 2015 Jan 5. PMID 25431345
- [Derived] Ruwald MH, Solomon SD, Foster E, Kutyifa V, Ruwald AC, Sherazi S, McNitt S, Jons C, Moss AJ, Zareba W. Left ventricular ejection fraction normalization in cardiac resynchronization therapy and risk of ventricular arrhythmias and clinical outcomes: results from the Multicenter Automatic Defibrillator Implantation Trial With Cardiac Resynchronization Therapy (MADIT-CRT) trial. Circulation. 2014 Dec 23;130(25):2278-86. doi: 10.1161/CIRCULATIONAHA.114.011283. Epub 2014 Oct 9. PMID 25301831
- [Derived] Ruwald MH, Mittal S, Ruwald AC, Aktas MK, Daubert JP, McNitt S, Al-Ahmad A, Jons C, Kutyifa V, Steinberg JS, Wang P, Moss AJ, Zareba W. Association between frequency of atrial and ventricular ectopic beats and biventricular pacing percentage and outcomes in patients with cardiac resynchronization therapy. J Am Coll Cardiol. 2014 Sep 9;64(10):971-81. doi: 10.1016/j.jacc.2014.06.1177. PMID 25190230
- [Derived] Ruwald AC, Kutyifa V, Ruwald MH, Solomon S, Daubert JP, Jons C, Brenyo A, McNitt S, Do D, Tanabe K, Al-Ahmad A, Wang P, Moss AJ, Zareba W. The association between biventricular pacing and cardiac resynchronization therapy-defibrillator efficacy when compared with implantable cardioverter defibrillator on outcomes and reverse remodelling. Eur Heart J. 2015 Feb 14;36(7):440-8. doi: 10.1093/eurheartj/ehu294. Epub 2014 Aug 11. PMID 25112662
- [Derived] Kutyifa V, Stockburger M, Daubert JP, Holmqvist F, Olshansky B, Schuger C, Klein H, Goldenberg I, Brenyo A, McNitt S, Merkely B, Zareba W, Moss AJ. PR interval identifies clinical response in patients with non-left bundle branch block: a Multicenter Automatic Defibrillator Implantation Trial-Cardiac Resynchronization Therapy substudy. Circ Arrhythm Electrophysiol. 2014 Aug;7(4):645-51. doi: 10.1161/CIRCEP.113.001299. Epub 2014 Jun 24. PMID 24963007
- [Derived] Brenyo A, Barsheshet A, Kutyifa V, Ruwald AC, Rao M, Zareba W, Pouleur AC, Knappe D, Solomon SD, McNitt S, Huang DT, Moss AJ, Goldenberg I. Predictors of spontaneous reverse remodeling in mild heart failure patients with left ventricular dysfunction. Circ Heart Fail. 2014 Jul;7(4):565-72. doi: 10.1161/CIRCHEARTFAILURE.113.000929. Epub 2014 Apr 30. PMID 24786217
- [Derived] Goldenberg I, Kutyifa V, Klein HU, Cannom DS, Brown MW, Dan A, Daubert JP, Estes NA 3rd, Foster E, Greenberg H, Kautzner J, Klempfner R, Kuniss M, Merkely B, Pfeffer MA, Quesada A, Viskin S, McNitt S, Polonsky B, Ghanem A, Solomon SD, Wilber D, Zareba W, Moss AJ. Survival with cardiac-resynchronization therapy in mild heart failure. N Engl J Med. 2014 May 1;370(18):1694-701. doi: 10.1056/NEJMoa1401426. Epub 2014 Mar 30. PMID 24678999
- [Derived] Ge Y, Ruwald AC, Kutyifa V, McNitt S, Polonsky S, Klein H, Goldenberg I, Solomon SD, Foster E, Zareba W, Moss AJ. A metric for evaluating the cardiac response to resynchronization therapy. Am J Cardiol. 2014 Apr 15;113(8):1371-7. doi: 10.1016/j.amjcard.2014.01.410. Epub 2014 Jan 31. PMID 24607029
- [Derived] Slyngstad T, Huth Ruwald AC, Kutyifa V, McNitt S, Polonsky B, Solomon SD, Foster E, Goldenberg I, Wang PJ, Klein H, Zareba W, Moss AJ. Cardiac resynchronization therapy is associated with reductions in left atrial volume and inappropriate implantable cardioverter-defibrillator therapy in MADIT-CRT. Heart Rhythm. 2014 Jun;11(6):1001-7. doi: 10.1016/j.hrthm.2014.01.033. Epub 2014 Feb 4. PMID 24502968
- [Derived] Kuperstein R, Goldenberg I, Moss AJ, Solomon S, Bourgoun M, Shah A, McNitt S, Zareba W, Klempfner R. Left atrial volume and the benefit of cardiac resynchronization therapy in the MADIT-CRT trial. Circ Heart Fail. 2014 Jan;7(1):154-60. doi: 10.1161/CIRCHEARTFAILURE.113.000748. Epub 2013 Dec 17. PMID 24347664
- [Derived] Ruwald AC, Pietrasik G, Goldenberg I, Kutyifa V, Daubert JP, Ruwald MH, Jons C, McNitt S, Wang P, Zareba W, Moss AJ. The effect of intermittent atrial tachyarrhythmia on heart failure or death in cardiac resynchronization therapy with defibrillator versus implantable cardioverter-defibrillator patients: a MADIT-CRT substudy (Multicenter Automatic Defibrillator Implantation Trial With Cardiac Resynchronization Therapy). J Am Coll Cardiol. 2014 Apr 1;63(12):1190-1197. doi: 10.1016/j.jacc.2013.10.074. Epub 2013 Dec 11. PMID 24333490
- [Derived] Sood N, Ruwald AC, Solomon S, Daubert JP, McNitt S, Polonsky B, Jons C, Clyne CA, Zareba W, Moss AJ. Association between myocardial substrate, implantable cardioverter defibrillator shocks and mortality in MADIT-CRT. Eur Heart J. 2014 Jan;35(2):106-15. doi: 10.1093/eurheartj/eht451. Epub 2013 Oct 31. PMID 24179073
- [Derived] Brenyo A, Barsheshet A, Rao M, Huang DT, Zareba W, McNitt S, Hall WJ, Peterson DR, Solomon SD, Moss AJ, Goldenberg I. Brain natriuretic peptide and cardiac resynchronization therapy in patients with mildly symptomatic heart failure. Circ Heart Fail. 2013 Sep 1;6(5):998-1004. doi: 10.1161/CIRCHEARTFAILURE.112.000174. Epub 2013 Jun 25. PMID 23801020
- [Derived] Ruwald MH, Abu-Zeitone A, Jons C, Ruwald AC, McNitt S, Kutyifa V, Zareba W, Moss AJ. Impact of carvedilol and metoprolol on inappropriate implantable cardioverter-defibrillator therapy: the MADIT-CRT trial (Multicenter Automatic Defibrillator Implantation With Cardiac Resynchronization Therapy). J Am Coll Cardiol. 2013 Oct 8;62(15):1343-50. doi: 10.1016/j.jacc.2013.03.087. Epub 2013 Jun 13. PMID 23770172
- [Derived] Kutyifa V, Pouleur AC, Knappe D, Al-Ahmad A, Gibinski M, Wang PJ, McNitt S, Merkely B, Goldenberg I, Solomon SD, Moss AJ, Zareba W. Dyssynchrony and the risk of ventricular arrhythmias. JACC Cardiovasc Imaging. 2013 Apr;6(4):432-44. doi: 10.1016/j.jcmg.2012.12.008. PMID 23579010
- [Derived] Ruwald MH, Ruwald AC, Jons C, Alexis J, McNitt S, Zareba W, Moss AJ. Effect of metoprolol versus carvedilol on outcomes in MADIT-CRT (multicenter automatic defibrillator implantation trial with cardiac resynchronization therapy). J Am Coll Cardiol. 2013 Apr 9;61(14):1518-26. doi: 10.1016/j.jacc.2013.01.020. PMID 23500269
- [Derived] Kutyifa V, Kloppe A, Zareba W, Solomon SD, McNitt S, Polonsky S, Barsheshet A, Merkely B, Lemke B, Nagy VK, Moss AJ, Goldenberg I. The influence of left ventricular ejection fraction on the effectiveness of cardiac resynchronization therapy: MADIT-CRT (Multicenter Automatic Defibrillator Implantation Trial With Cardiac Resynchronization Therapy). J Am Coll Cardiol. 2013 Mar 5;61(9):936-44. doi: 10.1016/j.jacc.2012.11.051. PMID 23449428
- [Derived] Brenyo A, Rao M, Barsheshet A, Cannom D, Quesada A, McNitt S, Huang DT, Moss AJ, Zareba W. QRS axis and the benefit of cardiac resynchronization therapy in patients with mildly symptomatic heart failure enrolled in MADIT-CRT. J Cardiovasc Electrophysiol. 2013 Apr;24(4):442-8. doi: 10.1111/jce.12057. Epub 2012 Dec 17. PMID 23252875
- [Derived] Goldstein RE, Haigney MC, Krone RJ, McNitt S, Zareba W, Moss AJ. Differing effects of cardiac resynchronization therapy on long-term mortality in patient subgroups of MADIT-CRT defined by baseline conduction and 1-year post-treatment left ventricular remodeling. Heart Rhythm. 2013 Mar;10(3):366-73. doi: 10.1016/j.hrthm.2012.11.020. Epub 2012 Nov 24. PMID 23183194
- [Derived] Ouellet G, Huang DT, Moss AJ, Hall WJ, Barsheshet A, McNitt S, Klein H, Zareba W, Goldenberg I. Effect of cardiac resynchronization therapy on the risk of first and recurrent ventricular tachyarrhythmic events in MADIT-CRT. J Am Coll Cardiol. 2012 Oct 30;60(18):1809-16. doi: 10.1016/j.jacc.2012.05.057. Epub 2012 Oct 3. PMID 23040580
- [Derived] Hsu JC, Solomon SD, Bourgoun M, McNitt S, Goldenberg I, Klein H, Moss AJ, Foster E; MADIT-CRT Executive Committee. Predictors of super-response to cardiac resynchronization therapy and associated improvement in clinical outcome: the MADIT-CRT (multicenter automatic defibrillator implantation trial with cardiac resynchronization therapy) study. J Am Coll Cardiol. 2012 Jun 19;59(25):2366-73. doi: 10.1016/j.jacc.2012.01.065. PMID 22698490
- [Derived] Brenyo A, Link MS, Barsheshet A, Moss AJ, Zareba W, Wang PJ, McNitt S, Huang D, Foster E, Estes M 3rd, Solomon SD, Goldenberg I. Cardiac resynchronization therapy reduces left atrial volume and the risk of atrial tachyarrhythmias in MADIT-CRT (Multicenter Automatic Defibrillator Implantation Trial with Cardiac Resynchronization Therapy). J Am Coll Cardiol. 2011 Oct 11;58(16):1682-9. doi: 10.1016/j.jacc.2011.07.020. PMID 21982313
- [Derived] Goldenberg I, Moss AJ, Hall WJ, Foster E, Goldberger JJ, Santucci P, Shinn T, Solomon S, Steinberg JS, Wilber D, Barsheshet A, McNitt S, Zareba W, Klein H; MADIT-CRT Executive Committee. Predictors of response to cardiac resynchronization therapy in the Multicenter Automatic Defibrillator Implantation Trial with Cardiac Resynchronization Therapy (MADIT-CRT). Circulation. 2011 Oct 4;124(14):1527-36. doi: 10.1161/CIRCULATIONAHA.110.014324. Epub 2011 Sep 6. PMID 21900084
- [Derived] Goldenberg I, Hall WJ, Beck CA, Moss AJ, Barsheshet A, McNitt S, Polonsky S, Brown MW, Zareba W. Reduction of the risk of recurring heart failure events with cardiac resynchronization therapy: MADIT-CRT (Multicenter Automatic Defibrillator Implantation Trial With Cardiac Resynchronization Therapy). J Am Coll Cardiol. 2011 Aug 9;58(7):729-37. doi: 10.1016/j.jacc.2011.04.024. PMID 21816309
- [Derived] Barsheshet A, Wang PJ, Moss AJ, Solomon SD, Al-Ahmad A, McNitt S, Foster E, Huang DT, Klein HU, Zareba W, Eldar M, Goldenberg I. Reverse remodeling and the risk of ventricular tachyarrhythmias in the MADIT-CRT (Multicenter Automatic Defibrillator Implantation Trial-Cardiac Resynchronization Therapy). J Am Coll Cardiol. 2011 Jun 14;57(24):2416-23. doi: 10.1016/j.jacc.2010.12.041. PMID 21658562
- [Derived] Knappe D, Pouleur AC, Shah AM, Cheng S, Uno H, Hall WJ, Bourgoun M, Foster E, Zareba W, Goldenberg I, McNitt S, Pfeffer MA, Moss AJ, Solomon SD; Multicenter Automatic Defibrillator Implantation Trial-Cardiac Resynchronization Therapy Investigators. Dyssynchrony, contractile function, and response to cardiac resynchronization therapy. Circ Heart Fail. 2011 Jul;4(4):433-40. doi: 10.1161/CIRCHEARTFAILURE.111.962902. Epub 2011 May 22. PMID 21602574
- [Derived] Singh JP, Klein HU, Huang DT, Reek S, Kuniss M, Quesada A, Barsheshet A, Cannom D, Goldenberg I, McNitt S, Daubert JP, Zareba W, Moss AJ. Left ventricular lead position and clinical outcome in the multicenter automatic defibrillator implantation trial-cardiac resynchronization therapy (MADIT-CRT) trial. Circulation. 2011 Mar 22;123(11):1159-66. doi: 10.1161/CIRCULATIONAHA.110.000646. Epub 2011 Mar 7. PMID 21382893
- [Derived] Zareba W, Klein H, Cygankiewicz I, Hall WJ, McNitt S, Brown M, Cannom D, Daubert JP, Eldar M, Gold MR, Goldberger JJ, Goldenberg I, Lichstein E, Pitschner H, Rashtian M, Solomon S, Viskin S, Wang P, Moss AJ; MADIT-CRT Investigators. Effectiveness of Cardiac Resynchronization Therapy by QRS Morphology in the Multicenter Automatic Defibrillator Implantation Trial-Cardiac Resynchronization Therapy (MADIT-CRT). Circulation. 2011 Mar 15;123(10):1061-72. doi: 10.1161/CIRCULATIONAHA.110.960898. Epub 2011 Feb 28. PMID 21357819
- [Derived] Martin DT, McNitt S, Nesto RW, Rutter MK, Moss AJ. Cardiac resynchronization therapy reduces the risk of cardiac events in patients with diabetes enrolled in the multicenter automatic defibrillator implantation trial with cardiac resynchronization therapy (MADIT-CRT). Circ Heart Fail. 2011 May;4(3):332-8. doi: 10.1161/CIRCHEARTFAILURE.110.959510. Epub 2011 Feb 24. PMID 21350054
- [Derived] Arshad A, Moss AJ, Foster E, Padeletti L, Barsheshet A, Goldenberg I, Greenberg H, Hall WJ, McNitt S, Zareba W, Solomon S, Steinberg JS; MADIT-CRT Executive Committee. Cardiac resynchronization therapy is more effective in women than in men: the MADIT-CRT (Multicenter Automatic Defibrillator Implantation Trial with Cardiac Resynchronization Therapy) trial. J Am Coll Cardiol. 2011 Feb 15;57(7):813-20. doi: 10.1016/j.jacc.2010.06.061. PMID 21310317
- [Derived] Solomon SD, Foster E, Bourgoun M, Shah A, Viloria E, Brown MW, Hall WJ, Pfeffer MA, Moss AJ; MADIT-CRT Investigators. Effect of cardiac resynchronization therapy on reverse remodeling and relation to outcome: multicenter automatic defibrillator implantation trial: cardiac resynchronization therapy. Circulation. 2010 Sep 7;122(10):985-92. doi: 10.1161/CIRCULATIONAHA.110.955039. Epub 2010 Aug 23. PMID 20733097
- [Derived] Barsheshet A, Goldenberg I, Narins CR, Moss AJ, McNitt S, Wang PJ, Huang DT, Hall WJ, Zareba W, Eldar M, Guetta V. Time dependence of life-threatening ventricular tachyarrhythmias after coronary revascularization in MADIT-CRT. Heart Rhythm. 2010 Oct;7(10):1421-7. doi: 10.1016/j.hrthm.2010.07.005. Epub 2010 Jul 8. PMID 20620231
- [Derived] Moss AJ, Hall WJ, Cannom DS, Klein H, Brown MW, Daubert JP, Estes NA 3rd, Foster E, Greenberg H, Higgins SL, Pfeffer MA, Solomon SD, Wilber D, Zareba W; MADIT-CRT Trial Investigators. Cardiac-resynchronization therapy for the prevention of heart-failure events. N Engl J Med. 2009 Oct 1;361(14):1329-38. doi: 10.1056/NEJMoa0906431. Epub 2009 Sep 1. PMID 19723701

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled 1820 patients from 110 hospital centers (88 in the United States, 2 in Canada, and 20 in Europe) between December 22, 2004 and April 23, 2008. Follow-up continued thereafter until trial termination.
Pre-assignment Details: Data from all patients enrolled were analyzed on an intention-to-treat basis.
Groups:
- Cardiac Resynchronization Therapy + Defibrillator: Patients randomized to cardiac resynchronization therapy with backup defibrillation (CRT-D) in addition to optimal pharmacologic therapy (as administered by the primary care physician). CRT-D devices both deliver shocks to terminate potentially lethal ventricular arrhythmias and pace both ventricles in patients with ventricular dyssynchrony.
- Implantable Cardioverter Defibrillator Alone: Patients randomized to implantable cardioverter defibrillator (ICD) in addition to optimal pharmacologic therapy (as administered by the primary care physician). ICDs deliver shocks to terminate potentially lethal ventricular arrhythmias.
Period: Overall Study
Arm/Group | Cardiac Resynchronization Therapy + Defibrillator | Implantable Cardioverter Defibrillator Alone
Started | 1089 | 731
Completed | 1089 | 731
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cardiac Resynchronization Therapy + Defibrillator | Implantable Cardioverter Defibrillator Alone | Total
Number analyzed (Participants) | 1089 | 731 | 1820
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 543 | 380 | 923
  >=65 years | 546 | 351 | 897
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (11) | 64 (11) | 65 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 275 | 178 | 453
  Male | 814 | 553 | 1367
Region of Enrollment [Number; unit: participants]
  United States | 757 | 514 | 1271
  Canada | 14 | 8 | 22
  Czech Republic | 17 | 11 | 28
  Denmark | 22 | 13 | 35
  France | 13 | 9 | 22
  Germany | 98 | 61 | 159
  Hungary | 16 | 10 | 26
  Israel | 45 | 30 | 75
  Italy | 15 | 12 | 27
  Netherlands | 34 | 24 | 58
  Poland | 14 | 10 | 24
  Spain | 36 | 24 | 60
  Switzerland | 4 | 2 | 6
  United Kingdom | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Mortality From Any Cause or First Heart Failure (HF) Event
Description: MADIT-CRT was an event-driven trial in which patients were monitored for all-cause mortality and HF events. An HF event was defined as either hospitalization for symptoms and/or signs consistent with congestive HF and:
  1. administration of intravenous decongestive therapy that does not involve formal in-patient hospital admission, regardless of the setting (i.e. in an emergency room setting, in the physician's office, etc.), or
  2. administration of an augmented HF regimen with oral or intravenous medications during an in-hospital stay.
Time Frame: Outcome measured at average follow-up duration of 2.4 years.
Population: Analysis was performed on an intention-to-treat basis and counted the time to first event. The category "Patients with Death at Any Time", includes deaths that occurred after the first heart failure event.
Measure: Number; unit: Participants
Arm/Group | Cardiac Resynchronization Therapy + Defibrillator | Implantable Cardioverter Defibrillator Alone
Number analyzed (Participants) | 1089 | 731
Participants
  Patients who are Event Free | 901 | 543
  Patients with Death or Heart Failure Event | 188 | 188
  Patients with Heart Failure Event Alone | 152 | 170
  Patients with Death at Any Time | 74 | 53
Statistical Analysis 1: Comparison: Cardiac Resynchronization Therapy + Defibrillator vs Implantable Cardioverter Defibrillator Alone; The trial utilized a Wang-Tsiatis (delta=0.1) group-sequential design with 95% power to detect a hazard ratio of 0.75 at a two-sided significance level of 0.05. Primary analysis based on statistical evaluation comparing the life-table event-free survival time graphs for CRT-D and ICD-only arms of the trial. Stratified Cox proportional-hazards regression was used to estimate a hazard ratio and statistical significance was evaluated with the log-rank test. Stratified by center and ischemic status; Test type: Superiority or Other; p < 0.001, Log Rank — The trial involved prespecified event monitoring at up to 20 successive periods by an independent DSMB to permit trial termination if the CRT-D was superior to, inferior to, or not different from ICD according to prespecified stopping rules; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.52 to 0.84] — A Hazard ratio < 1.0 would indicate that the result favors CRT-D

2. Secondary Outcome: Recurrent Heart Failure Events
Description: The MADIT-CRT secondary outcome evaluated the effects of CRT-D, relative to ICD, on the recurrence of heart failure events over the full study period An HF event was defined as either hospitalization for symptoms and/or signs consistent with congestive HF and:
  1. administration of intravenous decongestive therapy that does not involve formal in-patient hospital admission, regardless of the setting (i.e. in an emergency room setting, in the physician's office, etc.), or
  2. administration of an augmented HF regimen with oral or intravenous medications during an in-hospital stay.
Time Frame: Time of event, DSMB review
Measure: Count of Participants; unit: Participants
Groups:
- ICD: Implantable Cardioverter Defibrillator: ICD: Implantable cardioverter defibrillator
  Implantable Cardioverter Defibrillator (ICD): Boston Scientific Corporation Market Released Implantable Cardioverter Defibrillator
Arm/Group | CRT-D | ICD: Implantable Cardioverter Defibrillator
Number analyzed (Participants) | 1089 | 731
Participants
  Participants with 0 events | 928 | 545
  Participants with 1 event | 93 | 107
  Participants with 2 or more events | 68 | 79
Statistical Analysis 1: Comparison: CRT-D vs ICD: Implantable Cardioverter Defibrillator; Test type: Superiority; p = 0.001, Andersen-Gill; Andersen-Gill model performed, adjusted for a previous HF event in the study, stratified by ischemic status and using robust variance estimation; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.53 to 0.86] — Model adjusted for previously experienced heart failure event in the study. Hazard Ratio (95% CI) comparing patients with a previous heart failure event to those patients without a prior heart failure event equaled 8.84 (6084, 11.43), p<0.001

ADVERSE EVENTS:
Time Frame: 91 Days
Description: The primary outcome was performed on an intention-to-treat basis and all participants were followed. However, the number of participants at risk for adverse events is fewer than the total number in the primary outcome. Some participants did not undergo the surgical procedure for device implant and were therefore not subjected to risk.
Arm/Group | Cardiac Resynchronization Therapy + Defibrillator | Implantable Cardioverter Defibrillator Alone
Serious Adverse Events (participants affected / at risk) | 164/1079 | 55/712
Other Adverse Events (participants affected / at risk) | 126/1079 | 0/712
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cardiac Resynchronization Therapy + Defibrillator (N=1079) | Implantable Cardioverter Defibrillator Alone (N=712)
Lead Dislodgment, Left Ventricular (Cardiac disorders) | 46 (51) | 1 (1)
Lead Dislodgment, Right Atrial (Cardiac disorders) | 33 (33) | 10 (10)
Pneumothorax (Surgical and medical procedures) | 15 (15) | 5 (5)
Hematoma, Pocket (Surgical and medical procedures) | 14 (14) | 5 (5)
Extracardiac Stimulation, Left Ventricular (Cardiac disorders) | 11 (11) | 0 (0)
Lead Dislodgment, Right Ventricular (Cardiac disorders) | 8 (8) | 5 (5)
Thromboembolic Events (Blood and lymphatic system disorders) | 8 (8) | 4 (4)
Atrioventricular Block (Surgical and medical procedures) | 6 (6) | 2 (2)
Adverse Reaction (Surgical and medical procedures) | 6 (6) | 7 (7)
Elevated Threshold, Right Ventricular (Cardiac disorders) | 6 (6) | 3 (3)
Infection, Post Surgical (Surgical and medical procedures) | 9 (9) | 2 (2)
Inadvertent Ventricular Tachyarrhythmia (Cardiac disorders) | 4 (4) | 2 (2) — Arrhythmia inadvertently induced during implant procedure.
Renal Failure (Surgical and medical procedures) | 4 (4) | 0 (0) — Secondary to use of contrast media
Pericardial Effusion (Surgical and medical procedures) | 3 (4) | 1 (1)
Myocardial Perforation with Tamponade (Surgical and medical procedures) | 3 (3) | 1 (1)
Elevated Defibrillation Thresholds (Cardiac disorders) | 6 (6) | 8 (8)
Hemorrhage, Pocket (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Inappropriate Tachyarrhythmia Therapy (Cardiac disorders) | 2 (2) | 1 (1)
Early Elective Replacement Indicator (Cardiac disorders) | 2 (2) | 1 (1)
Insulation Breach, Left Ventricular Lead (Cardiac disorders) | 2 (2) | 0 (0)
Inadvertent Supraventricular Tachyarrhythmia (Cardiac disorders) | 2 (2) | 0 (0)
Arterial Perforation (Surgical and medical procedures) | 1 (1) | 0 (0)
Venous Occlusion (Surgical and medical procedures) | 1 (1) | 0 (0)
Seroma, Pocket (Surgical and medical procedures) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Worsening Heart Failure (Cardiac disorders) | 2 (2) | 1 (1)
Elevated Threshold, Left Ventricular (Cardiac disorders) | 1 (1) | 0 (0)
Difficulty Measing Impedance/Amplitude (Cardiac disorders) | 1 (1) | 0 (0)
Pulse Generator Migration (Surgical and medical procedures) | 1 (1) | 0 (0)
Set Screws Not Tightened (Surgical and medical procedures) | 0 (0) | 3 (3)
Post Surgical Wound Discomfort (Surgical and medical procedures) | 0 (0) | 1 (1)
Elevated Shock Impedance (Cardiac disorders) | 1 (1) | 0 (0)
Bigeminy (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cardiac Resynchronization Therapy + Defibrillator (N=1079) | Implantable Cardioverter Defibrillator Alone (N=712)
Extracardiac Stimulation, Left Ventricular (Cardiac disorders) | 70 (77) | 0 (0) — Events corrected non-invasively with reprogramming.
Pacemaker Mediated Tachycardia (Cardiac disorders) | 56 (67) | 0 (0) — Events corrected non-invasively with reprogramming.

LIMITATIONS AND CAVEATS:
The FDA Circulatory Devices advisory panel recommended approval for the patient subpopulation with left bundle branch block (LBBB) only. Consequently, FDA has restricted indications for use to LBBB.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No